CLINICAL TRIAL: NCT05958290
Title: Cardiac Implantable Electronic Device Lifelong Antibiotic thErapy vs Stop and See The CIEDLESS Study A Prospective Study
Brief Title: Cardiac Implantable Electronic Device Lifelong Antibiotic thErapy vs Stop and See
Acronym: CIEDLESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Emil Loldrup Fosbol, Professor, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-23029723
Record Dates: First submitted 2023-07-05; First posted 2023-07-24 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Cardiac Implantable Electronic Device Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Discontinuation of antibiotics (Experimental)
  Interventions: Other: Discontinuation of antibiotics
- Standard treatment (No Intervention)

INTERVENTIONS:
Other: Discontinuation of antibiotics — Discontinuation of antibiotic treatment after at least 10 days iv antibiotic therapy and then per oral treatment to at least 6 weeks total.
  Arms: Discontinuation of antibiotics

SUMMARY:
The goal of this non-randomized prospective study is to test whether 6-weeks antibiotic treatment can cure an cardiac implantable electronic device (CIED) infection in patients where device extraction is not feasible.

The main question it aims to answer:

• Is 6-weeks medical therapy effective in curing definite CIED infection with device retention?

Participants will discontinue the antibiotic treatment after at least 10 days iv antibiotic therapy and then per oral treatment to at least 6 weeks total. After discontinuation of antibiotics, patients are closely observed for bacterial relapse.

For patients who are not interested in participation and who do not have exclusion criteria, we will ask for consent into a registry as we wish to compare patients undergoing discontinuation of antibiotics with patients undergoing standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Definite CIED infection by the EHRA criteria
* Deemed non-eligible for CIED extraction

Exclusion Criteria:

* Unavailable for follow-up (e.g., tourist)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of death or relapse bacteremia | 12 months
  Composite endpoint of all-cause mortality or relapse bacteremia with the primary pathogen

SECONDARY OUTCOMES:
Death | 12 months
  All-cause mortality. The number of patients who die within 12 months will be assessed for the main study arm as well as the registry study arm through medical chart review.
Readmission for any cause | 12 months
  The number of patients readmitted for any cause will be examined for the main study arm as well as the registry study arm through medical chart review.
Device extraction | 12 months
  The number of patients who have their device extracted will be assessed for the main study arm as well as the registry study arm through medical chart review..
Change in quality of life | 12 months
  Quality of life will be assessed at inclusion and after 12 months using the Kansas City Cardiomyopathy Questionnaire (KCCQ) evaluated with a face-to-face interview. We will evaluate changes in KCCQ scores from inclusion to end of follow-up. This outcome will only be assessed for the main study arm.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No